CLINICAL TRIAL: NCT05033886
Title: A Phase 3b, Randomized, Double-blind, Placebo-controlled, 24-week Study to Assess the Efficacy and Safety of Fezolinetant in Menopausal Women Suffering From Moderate to Severe Vasomotor Symptoms (Hot Flashes) and Considered Unsuitable for Hormone Replacement Therapy
Brief Title: A Study of Fezolinetant to Treat Hot Flashes in Women Going Through Menopause
Acronym: Daylight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2693-CL-0312; 2021-001685-38 (EudraCT Number)
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Vasomotor Symptoms
Keywords: ESN364; menopause; fezolinetant; vasomotor symptoms
MeSH Terms: interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- fezolinetant (Experimental): Participants receive fezolinetant 45 milligrams (mg) (one 30 mg tablet and one 15 mg tablet) orally once daily for 24 weeks of treatment.
  Interventions: Drug: fezolinetant
- placebo (Placebo Comparator): Participants receive placebo matched to fezolinetant tablets orally once daily for 24 weeks of treatment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fezolinetant — oral
  Other Names: ESN364
  Arms: fezolinetant
Drug: placebo — oral
  Arms: placebo

SUMMARY:
This study is for women in menopause who have moderate to severe hot flashes. It is for women who are unable to use hormone replacement therapy (HRT). Menopause, a normal part of life, is the time after a woman's last period. Hot flashes often occur during menopause. They can disrupt a woman's daily life.

The study medicines (also called investigational products, or IP) are tablets of fezolinetant or placebo. An investigational product means that the product is not yet licensed. In this study, a placebo is a dummy treatment that looks like fezolinetant but does not have any medicine in it. The study will compare fezolinetant with the placebo to learn if fezolinetant reduces the number and severity of hot flashes.

Women that want to take part in the study will be given an electronic handheld device with an app to track their hot flashes. Some women may be able to use the app on their own smartphone. In the last 10 days before their next clinic visit, the women will record information about their hot flashes. They can take part in the study if they have an average of 7 or more moderate to severe hot flashes each day. Women will be picked for 1 of 2 treatments (fezolinetant or placebo) by chance alone.

Women who take part in the study will take 2 tablets every day for 24 weeks. Treatment will be double-blinded. That means that the women in the study and the study doctors will not know who takes which of the study medicines (fezolinetant or placebo). The women will continue recording information about their hot flashes on the electronic device or their phone. They will also use another device to answer questions about how hot flashes affect their daily life.

During the study, the women will visit their study clinic several times for a check-up. This will happen during Weeks 2, 4, 8, 12, 16, 20, 24, and 27. Some women may be able to have home visits instead, from Week 2 to Week 20. At the check-up, they will be asked if they have any medical problems. Other checks will include vital signs (heart rate, temperature and blood pressure) and some blood samples taken for laboratory tests. At some check-ups, the women will have a physical exam. In Week 2 and Week 24, the women will have an ECG to check their heart rhythm. Women who have a uterus will also have a test called a transvaginal ultrasound. A probe is gently placed inside the vagina. Sound waves will create a picture of the organs in the pelvis. This will allow the study doctor to look more closely at the uterus and surrounding organs.

The last check-up (at Week 27) will be 3 weeks after they take their last tablets of study medicine (fezolinetant or placebo).

ELIGIBILITY:
Inclusion Criteria :

* Participant must be seeking treatment or relief for vasomotor symptoms (VMS) associated with menopause and confirmed as menopausal per one of the following criteria at the screening visit:

  * Spontaneous amenorrhea for >= 12 consecutive months
  * Spontaneous amenorrhea for >= 6 months with biochemical criterion of menopause (follicle-stimulating hormone [FSH] > 40 IU/L)
  * Had bilateral oophorectomy >= 6 weeks prior to the screening visit (with or without hysterectomy)
* Participant has VMS and is unsuitable to receive hormone replacement therapy (HRT) (HRT contraindicated, HRT caution, HRT stoppers and HRT averse participants).
* Participant has a minimum average of 7 moderate to severe hot flash's (HFs) (VMS) per day as recorded in the electronic diary during the last 10 days prior to randomization.
* Participant is in good general health as determined on the basis of medical history, general physical examination, laboratory and other medical assessments.
* Participant has a negative serology panel (including hepatitis B surface antigen, hepatitis C virus antibody and human immunodeficiency virus antibody screens).
* Had hysterectomy without oophorectomy and who meets the biochemical criterion of menopause (FSH > 40 IU/L).

Exclusion Criteria:

* Participant uses a prohibited therapy for VMS (e.g., prescription, over-the-counter or herbal) prior to screening and for the duration of treatment with investigational product (IP).
* Participant has known documented substance abuse or alcohol addiction within 6 months of screening.
* Participant has history of a malignant tumor within the last 5 years, except for basal cell carcinoma.
* Participant has endometrial thickness > 8 mm on the locally read screening transvaginal ultrasound (TVU) or any clinically significant findings that that would make the participant ineligible.
* Participant has history of severe allergy, hypersensitivity or intolerance to the IP and/or any of its excipients.
* Participant has a history of seizures or other convulsive disorders unless well controlled.
* Participant has a medical condition or chronic disease (including history of neurological [including cognitive], renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Participant has any of the following: active liver disease, jaundice, elevated liver aminotransferases at screening (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]), elevated total bilirubin (TBL) or direct bilirubin (DBL) > 1.5 × upper limit of normal (ULN), elevated International Normalized Ratio (INR) > 1.5 (unless participant is receiving anticoagulant therapy) or elevated alkaline phosphatase (ALP). Participants with mildly elevated ALT or AST up to 1.5 × ULN can be enrolled if TBL and DBL are normal. Participants with mildly elevated ALP (up to 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Participants with Gilbert's syndrome with elevated TBL may be enrolled as long as DBL, hemoglobin and reticulocytes are normal.
* Participant has creatinine > 1.5 × ULN or estimated glomerular filtration rate using the Modification of Diet in Renal Disease formula <= 59 mL/min per 1.73 m^2 at the screening visit.
* Participant has a history of suicide attempt or suicidal behavior within the last 12 months.
* Participant has participated in another interventional study within the last 30 days prior to screening and for the duration of the study.
* Participant who has been previously enrolled in a clinical study with fezolinetant.
* Participant is unable or unwilling to complete the study procedures.
* Participant has any condition makes the participant unsuitable for study participation.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Mean change in the frequency of moderate to severe VMS from baseline at week 24 | Baseline, week 24
  The frequency of moderate to severe VMS is the number of moderate to severe VMS per 24 hours. A daily frequency per week is derived by taking the mean of the data over 7 days. Moderate VMS is defined as sensation of heat with sweating/dampness but is able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity.

SECONDARY OUTCOMES:
Mean change in the severity of moderate to severe VMS from baseline at week 24 | Baseline, week 24
  Severity of moderate to severe VMS per day is calculated as follows: [(number of moderate Hot Flashes (HFs) × 2) + (number of severe HFs/day × 3)]/number of daily moderate/severe HFs. Moderate VMS is defined as sensation of heat with sweating but able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, causing cessation of activity. Severity is zero for participants that have had no moderate or severe VMS. Higher score indicates greater severity. A negative change indicates a reduction/improvement.
Mean change in the patient-reported sleep disturbance by the Patient-reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8b (PROMIS SD SF 8b total score) from baseline at week 24 | Baseline, week 24
  The PROMIS SD SF 8b assesses self reported sleep disturbance over the past 7 days and includes perceptions of restless sleep; satisfaction with sleep; refreshing sleep; difficulties sleeping, getting to sleep or staying asleep; amount of sleep; and sleep quality. Because it assesses the participants experience of sleep disturbance, the measure does not focus on specific sleep-disorder symptoms or ask participants to report objective measures of sleep (e.g., total amount of sleep, time to fall asleep and amount of wakefulness during sleep). Responses to each of the 8 items range from 1 (no disturbed sleep) to 5 (disturbed sleep), and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS SD SF 8b indicate more of the disturbed sleep. A negative value indicates a better outcome.
Mean change in the frequency of moderate to severe VMS from baseline at weeks 1, 4, 8, 12, 16 and 20 | Baseline, weeks 1, 4, 8, 12, 16 and 20
  The frequency of moderate to severe VMS is the number of moderate to severe VMS per 24 hours. A daily frequency per week is derived by taking the mean of the data over 7 days. Moderate VMS is defined as sensation of heat with sweating/dampness but is able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity.
Mean change in severity of moderate to severe VMS from baseline at weeks 1, 4, 8, 12, 16 and 20 | Baseline, weeks 1, 4, 8, 12, 16 and 20
  Severity of moderate to severe VMS per day is calculated as follows: [(number of moderate HFs × 2) + (number of severe HFs/day × 3)]/number of daily moderate/severe HFs. Moderate VMS is defined as sensation of heat with sweating/dampness but is able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, causing cessation of activity. Severity is zero for participants that have had no moderate or severe VMS. Higher score indicates greater severity. A negative change indicates a reduction/improvement.
Mean percent change in the frequency of moderate to severe VMS from baseline at weeks 1, 4, 8, 12, 16, 20 and 24 | Baseline, weeks 1, 4, 8, 12, 16, 20 and 24
  The frequency of moderate to severe VMS is the number of moderate to severe VMS per 24 hours. A daily frequency per week is derived by taking the mean of the data over 7 days. Moderate VMS is defined as sensation of heat with sweating/dampness but is able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity.
Number of participants with percent reduction of >/= 50% in the frequency of moderate to severe VMS from baseline at weeks 1, 4, 8, 12, 16, 20 and 24 | Baseline, weeks 1, 4, 8, 12, 16, 20 and 24
  The frequency of moderate to severe VMS is the number of moderate to severe VMS per 24 hours. A daily frequency per week is derived by taking the mean of the data over 7 days. Moderate VMS is defined as sensation of heat with sweating/dampness but is able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity.
Number of participants with percent reduction of >/= 75% in the frequency of moderate to severe VMS from baseline at weeks 1, 4, 8, 12, 16, 20 and 24 | Baseline, weeks 1, 4, 8, 12, 16, 20 and 24
  The frequency of moderate to severe VMS is the number of moderate to severe VMS per 24 hours. A daily frequency per week is derived by taking the mean of the data over 7 days. Moderate VMS is defined as sensation of heat with sweating/dampness but is able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity.
Number of participants with percent reduction at 100% in the frequency of moderate to severe VMS from baseline at weeks 1, 4, 8, 12, 16, 20 and 24 | Baseline, weeks 1, 4, 8, 12, 16, 20 and 24
  The frequency of moderate to severe VMS is the number of moderate to severe VMS per 24 hours. A daily frequency per week is derived by taking the mean of the data over 7 days. Moderate VMS is defined as sensation of heat with sweating/dampness but is able to continue activity. Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity.
Number of participants with Treatment Emergent Adverse Events (TEAEs) | From first dose to week 27
  An AE is any untoward medical occurrence in a participant administered a study drug, which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable & unintended sign, symptom, or disease temporally associated with the use of medicinal product (MP) whether considered related to MP. A TEAE was defined as an AE observed after starting administration of study intervention and up to 21 days after the last dose of study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (69):
- Site BE32005, Tienen, Vlaams Brabant, Belgium
- Canada (11):
  - Site CA15008, Brampton, Ontario
  - Site CA15010, London, Ontario
  - Site CA15003, Sarnia, Ontario
  - Site CA15012, Montreal, Quebec
  - Site CA15014, Québec, Quebec
  - Site CA15011, Saint Charles Borromeee, Quebec
  - Site CA15001, Sherbrooke, Quebec
  - Site CA15005, Victoriaville, Quebec
  - Site CA15002, Québec
  - Site CA15009, Québec
  - Site CA15007, Québec
- Czechia (10):
  - Site CZ42007, Tábor, Jihočeský kraj
  - Site CZ42002, Vodňany, Jihočeský kraj
  - Site CZ42008, Brno
  - Site CZ42005, Cheb
  - Site CZ42010, České Budějovice
  - Site CZ42009, Hradec Králové
  - Site CZ42011, Náchod
  - Site CZ42003, Olomouc
  - Site CZ42004, Písek
  - Site CZ42006, Prague
- Denmark (4):
  - Site DK45003, Gandrup, North Denmark
  - Site DK45002, Odense, Region Syddanmark
  - Site DK45004, Vejle, Region Syddanmark
  - Site DK45005, Arhus C
- Finland (2):
  - Site FI35801, Kuopio
  - Site FI35803, Oulu
- France (2):
  - Site FR33003, La Rochelle
  - Site FR33001, Nantes
- Germany (5):
  - Site DE49004, Hamburg
  - Site DE49005, Hamburg
  - Site DE49002, Leipzig
  - Site DE49008, Muechen
  - Site DE49006, Schwerin
- Hungary (3):
  - Site HU36002, Debrecen
  - Site HU36004, Kecskemét
  - Site HU36001, Szekesfeherver
- Italy (2):
  - Site IT39002, Bologna
  - Site IT39006, Pavia
- Netherlands (2):
  - Site NL31001, Beek, Limburg
  - Site NL31004, Rotterdam
- Site NO47001, Hamar, Norway
- Poland (11):
  - Site PL48001, Szczecin, West Pomeranian Voivodeship
  - Site PL48003, Bialystok
  - Site PL48013, Bydgoszcz
  - Site PL48006, Katowice
  - Site PL48011, Katowice
  - Site PL48004, Katowice
  - Site PL48007, Lublin
  - Site PL48009, Siedice
  - Site PL48017, Skierniewice
  - Site PL48012, Skorzewo
  - Site PL48010, Zamość
- Spain (4):
  - Site ES34002, Alcobendas
  - Site ES34005, Centellas
  - Site ES34003, Leganés
  - Site ES34001, Madrid
- Sweden (3):
  - Site SE46004, Qerebro
  - Site SE46003, Stockholm
  - Site SE46002, Uppsala
- Turkey (Türkiye) (3):
  - Site TR90002, Konak, İzmir
  - Site TR90001, Ankara, Mamak
  - Site TR90008, Izmir
- United Kingdom (5):
  - Site GB44007, Corby, Northamptonshire
  - Site GB44004, Shipley, Yorkshire
  - Site GB44002, Coventry
  - Site GB44006, Northwood
  - Site GB44003, Orpington

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Schaudig K, Wang X, Bouchard C, Hirschberg AL, Cano A, Shapiro C M M, Stute P, Wu X, Miyazaki K, Scrine L, Nappi RE. Efficacy and safety of fezolinetant for moderate-severe vasomotor symptoms associated with menopause in individuals unsuitable for hormone therapy: phase 3b randomised controlled trial. BMJ. 2024 Nov 18;387:e079525. doi: 10.1136/bmj-2024-079525. PMID 39557487
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14505&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/2693-CL-0312/